CLINICAL TRIAL: NCT01197911
Title: The Effect of Hepatic Impairment on the Pharmacokinetics of Aleglitazar: A Multiple-centre, Open-label Study Following a Single Oral Dose of Aleglitazar to Subjects With Mild or Moderate Hepatic Impairment and Healthy Subjects With Normal Hepatic Function.
Brief Title: A Study of The Effect of Hepatic Impairment on The Pharmacokinetics of Aleglitazar
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: BP25240
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — aleglitazar

ARMS (3):
- Mild impairment (Experimental)
  Interventions: Drug: aleglitazar
- Moderate impairment (Experimental)
  Interventions: Drug: aleglitazar
- Normal HF (Experimental)
  Interventions: Drug: aleglitazar

INTERVENTIONS:
Drug: aleglitazar — single oral dose

SUMMARY:
This open-label study will assess the effects of hepatic impairment on the pharmacokinetics of a single oral dose of aleglitazar in subjects with mild or moderate hepatic impairment (Child-Pugh class A or B) and in matched control subjects with normal hepatic function. Subjects will receive a single oral dose of aleglitazar, with assessment of the pharmacokinetics of aleglitazar on Days 1-5. Anticipated duration of study for each enrolled subject is approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults, 18-70 years of age inclusive
* Normal hepatic function or mild to moderate impaired liver function (Child-Pugh class A or B)
* Body mass index (BMI) 18 to 40 kg/m2 inclusive
* Females must be either surgically sterile, postmenopausal, or willing to use two reliable methods of contraception for the duration of the study and started 3 months before study start

Exclusion Criteria:

* For subjects with hepatic impairment: evidence of progressive liver disease within the last 4 weeks, or biliary liver cirrhosis or other causes of hepatic impairment not related to parenchymal disorder and/or disease
* For healthy volunteers: positive test for hepatitis B or C, alcohol intake of more than 14 units per week, or history of clinically significant alcohol or drug abuse
* Acute infection or current malignancy requiring treatment
* History of clinically significant allergic disease or drug hypersensitivity
* Positive test for HIV-1 or HIV-2 at screening
* Participation in a clinical study with an investigational drug or new chemical entity within 2 months prior to screening
* Females who are pregnant or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Orlando, Florida
  - Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 38 participants with normal hepatic function, or with mild or moderate hepatic impairment were enrolled from 30 September 2010 to 05 August 2011 at 2 study sites in the U. S.
Groups:
- Normal Hepatic Function: Participants with normal hepatic function received a single oral dose of aleglitazar 150 microgram (mcg) tablet
- Mild Hepatic Impairment: Participants with mild hepatic impairment received a single oral dose of aleglitazar 150 mcg tablet
- Moderate Hepatic Impairment: Participants with moderate hepatic impairment received a single oral dose of aleglitazar 150 mcg tablet
Period: Overall Study
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Started | 18 | 10 | 10
Completed | 18 | 10 | 9
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Total
Number analyzed (Participants) | 18 | 10 | 10 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (5.36) | 46.7 (8.39) | 52.8 (6.14) | 49.3 (6.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 5 | 16
  Male | 10 | 7 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf) of Aleglitazar
Description: AUCinf was calculated by non-compartmental analysis using the linear trapezoidal rule, using relative actual time values.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72 and 96 hours post-dose
Population: The pharmacokinetics (PK) analysis population consisted of all participants who received the study drug and adhered to the protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (h)*nanogram (ng)/milliliter (mL)
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
hours (h)*nanogram (ng)/milliliter (mL) | 98.5 (27.2) | 113 (41.8) | 151 (29.6)
Statistical Analysis 1: Comparison: Normal Hepatic Function vs Mild Hepatic Impairment; This statistical analysis consisted of all evaluable hepatic impaired participants for whom at least one evaluable matching healthy participant was available; Test type: Superiority or Other; Geometric Least-Squares Mean Ratio = 1.1480, 90% CI 2-sided [0.9293 to 1.4182]
Statistical Analysis 2: Comparison: Normal Hepatic Function vs Moderate Hepatic Impairment; This statistical analysis consisted of all evaluable hepatic impaired participants for whom at least one evaluable matching healthy participant was available. One Participant with moderate hepatic impairment was not included in the statistical analysis of the PK parameters as there was no appropriate participant with normal hepatic function match; Test type: Superiority or Other; Geometric Least-Squares Mean Ratio = 1.5518, 90% CI 2-sided [1.2468 to 1.9314]

2. Secondary Outcome: AUCinf of M1 (RO4408754) and M6 (RO4583746)
Description: M1 and M6 are pharmacologically inactive metabolites of aleglitazar. AUCinf represents the area under the concentration-time curve of the analyte in plasma over the time interval from zero extrapolated to infinity. AUCinf was calculated by non-compartmental analysis using the linear trapezoidal rule, using relative actual time values.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72 and 96 hours post-dose
Population: The PK analysis population consisted of all participants who received the study drug and adhered to the protocol. Only participants with data available for specific metabolite were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
h*ng/mL
  M1 (n = 18, 9, 9) | 14.0 (32.9) | 17.1 (29.5) | 24.9 (22.4)
  M6 (n = 18, 10, 9) | 148 (27.8) | 169 (54.3) | 247 (35.2)

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Aleglitazar
Description: Cmax was obtained directly from the concentration-time data.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Normal Hepatic Function: Participants with normal hepatic function received a single oral dose of aleglitazar 150 mcg tablet
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
ng/mL | 21.2 (30.3) | 20.1 (25.8) | 22.1 (24.4)
Statistical Analysis 1: Comparison: Normal Hepatic Function vs Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric Least-Squares Mean Ratio = 0.9477, 90% CI 2-sided [0.7908 to 1.1356]
Statistical Analysis 2: Comparison: Normal Hepatic Function vs Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Geometric Least-Squares Mean Ratio = 1.0782, 90% CI 2-sided [0.8941 to 1.3002]

4. Secondary Outcome: Cmax of M1 and M6
Description: M1 and M6 are pharmacologically inactive metabolites of aleglitazar. Cmax was obtained directly from the concentration-time data.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
ng/mL
  M1 (n=18, 9, 9) | 2.00 (25.7) | 2.01 (40.8) | 2.38 (27.1)
  M6 (n= 18, 10, 9) | 4.59 (24.5) | 4.05 (54.4) | 4.05 (19.7)

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 48 Hours Post-dose (AUC0-48) of Aleglitazar, M1, and M6
Description: M1 and M6 are pharmacologically inactive metabolites of aleglitazar. AUC0-48 was calculated by non-compartmental analysis using the linear trapezoidal rule, using relative actual time values.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
h*ng/mL
  Aleglitazar (n = 18, 10, 10) | 97.3 (27.0) | 111 (39.6) | 149 (28.6)
  M1 (n = 18, 9, 9) | 13.8 (31.6) | 16.4 (29.5) | 24.0 (20.9)
  M6 (n = 18, 10, 9) | 112 (25.4) | 115 (52.7) | 137 (17.4)

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to the Last Quantifiable Time-point Post-dose (AUClast) of Aleglitazar, M1, and M6
Description: AUClast was calculated by non-compartmental analysis using the linear trapezoidal rule, using relative actual time values.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
h*ng/mL
  Aleglitazar (n= 18, 10, 10) | 97.5 (27.6) | 112 (41.6) | 150 (29.6)
  M1 (n= 18, 10, 10) | 12.5 (32.4) | 15.2 (29.6) | 22.3 (23.6)
  M6 (n= 18, 10, 10) | 137 (27.2) | 151 (52.0) | 186 (35.6)

7. Secondary Outcome: Apparent Total Body Clearance (CL/F) of Aleglitazar
Description: CL/F was calculated as dose/AUCinf, where AUCinf represents the area under the concentration-time curve of the analyte in plasma over the time interval from zero extrapolated to infinity.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72 and 96 hours post-dose
Population: The PK analysis population consisted of all participants who received the study drug and adhered to the protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
L/h | 1.52 (27.2) | 1.33 (41.8) | 0.990 (29.6)

8. Secondary Outcome: Renal Clearance (CLR) of Aleglitazar, M1, and M6
Description: CLR was calculated as Ae0-48/AUC0-48, where Ae0-48 as amount excreted in urine from time 0 to 48 hours post-dose and AUC0-48 represents area under the concentration-time curve of the analyte in plasma over the time interval from zero to the 48 hours post-dose.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72, and 96 hours post-dose for plasma; 0-4, 4-8, 8-12, 12-24, and 24-48 hours post-dose for urine
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
L/h
  Aleglitazar (n = 18, 10, 9) | NA (NA) — CLR of aleglitazar was not calculable since amount excreted in urine was below limit of quantification. | NA (NA) — CLR of aleglitazar was not calculable since amount excreted in urine was below limit of quantification. | NA (NA) — CLR of aleglitazar was not calculable since amount excreted in urine was below limit of quantification.
  M1 (n = 18, 9, 9) | 0.994 (68.5) | 1.26 (48.5) | 0.857 (46.6)
  M6 (n = 18, 10, 9) | 0.0427 (31.4) | 0.0565 (28.4) | 0.0454 (19.9)

9. Secondary Outcome: Apparent Non-renal Clearance (CLNR/F) of Aleglitazar
Description: Plasma and urine samples were collected for this PK parameter. CLNR/F was estimated as CL/F, based on the approximated formula of CLNR/F = (CL-CLR)/F with CLR of aleglitazar being equal to zero. CL/F was calculated as dose/AUCinf, where AUCinf represents the area under the concentration-time curve of the analyte in plasma over the time interval from zero extrapolated to infinity. CLR was calculated as Ae0-48/AUC0-48, where Ae0-48 as amount excreted in urine from time zero to 48 hours post-dose and AUC0-48 represents area under the concentration-time curve of the analyte in plasma over the time interval from zero to the 48 hours post-dose.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72 and 96 hours post-dose for plasma; 0-4, 4-8, 8-12, 12-24, and 24-48 hours post-dose for urine
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 9
L/h | 1.52 (27.2) | 1.33 (41.8) | 0.991 (31.5)

10. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Aleglitazar, M1, and M6
Description: M1 and M6 are pharmacologically inactive metabolites of aleglitazar. Tmax was measured as time to reach the maximum concentration in the plasma after post-dose.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72 and 96 hours post-dose
Population: The PK analysis population consisted of all participants who received the study drug and adhered to the protocol.
Measure: Mean (Full Range); unit: h
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
h
  Aleglitazar | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 3.00] | 1.00 [0.50 to 2.00]
  M1 | 2.01 [1.00 to 5.00] | 3.50 [2.00 to 5.00] | 4.00 [2.00 to 5.00]
  M6 | 9.00 [5.00 to 12.0] | 9.00 [5.00 to 15.0] | 24.0 [9.00 to 24.0]

11. Secondary Outcome: Apparent Terminal Half-life (t½) of Aleglitazar, M1, and M6
Description: M1 and M6 are pharmacologically inactive metabolites of aleglitazar. T1/2 is the time required for a given drug concentration in the plasma to decrease by 50%.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
h
  Aleglitazar (n = 18, 10, 10) | 7.59 (31.3) | 8.18 (29.1) | 8.04 (19.3)
  M1 (n = 18, 9, 9) | 6.11 (55.0) | 7.79 (57.4) | 9.37 (31.7)
  M6 (n = 18, 10, 9) | 25.6 (17.4) | 27.1 (19.4) | 35.1 (28.4)

12. Secondary Outcome: Elimination Rate Constant (Kel) of Aleglitazar
Description: The kel is fraction of a substance that is removed per unit time measured at any particular instant. It was calculated using at least 3 concentration-time points and ideally covered more than 2 half-lives.
Time Frame: 0-4, 4-8, 8-12, 12-24, and 24-48 hours post-dose
Population: The PK analysis population consisted of all participants who received the study drug and adhered to the protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
1/h | 0.0914 (31.3) | 0.0847 (29.1) | 0.0862 (19.3)

13. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Aleglitazar
Description: Vz/F is the apparent volume of distribution during terminal phase after non-intravenous administration. It was calculated as CL/F/kel, where CL/F was calculated as dose/AUCinf, where AUCinf represents the area under the concentration-time curve of the analyte in plasma over the time interval from zero extrapolated to infinity and kel as constant elimination rate of aleglitazar.
Time Frame: as for outcome 9
Population: The PK analysis population consisted of all participants who received the study drug and adhered to the protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
L | 16.7 (30.7) | 15.7 (22.5) | 11.5 (17.0)

14. Secondary Outcome: Amount Excreted in Urine From Time 0 to 48 Hours Post-dose (Ae0-48) of Aleglitazar, M1, and M6
Description: The cumulative amount excreted in urine Ae0-48 over the entire collection interval of 48 hours was calculated by adding the Ae of the intervals 0-4, 4-8, 8-12, 12-24, and 24-48 hours, where Ae was calculated by multiplying the urine volume within the collection interval by the associated drug concentration.
Time Frame: 0-4, 4-8, 8-12, 12-24, and 24-48 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
mcg
  Aleglitazar (n = 18, 10, 9) | NA (NA) — Ae0-48 of aleglitazar was not calculable since amount excreted in urine was below limit of quantification. | NA (NA) — Ae0-48 of aleglitazar was not calculable since amount excreted in urine was below limit of quantification. | NA (NA) — Ae0-48 of aleglitazar was not calculable since amount excreted in urine was below limit of quantification.
  M1 (n = 18, 10, 10) | 13.7 (49.1) | 21.1 (31.8) | 20.5 (47.0)
  M6 (n = 18, 10, 10) | 4.78 (39.7) | 6.48 (53.2) | 5.81 (37.3)

15. Secondary Outcome: Fraction of Drug Excreted in Urine From Time 0 to 48 Hours Post-dose (fe0-48) of Aleglitazar
Description: fe0-48 was calculated as Ae0-48/dose. The cumulative amount excreted in urine Ae0-48 over the entire collection interval of 48 hours was calculated by adding the Ae of the intervals 0-4, 4-8, 8-12, 12-24, and 24-48 hours. Ae was calculated by multiplying the urine volume within the collection interval by the associated drug concentration.
Time Frame: 0-4, 4-8, 8-12, 12-24, and 24-48 hours post-dose
Population: The PK analysis population consisted of all participants who received the study drug and adhered to the protocol. Only participants with data available for specific metabolite were analyzed. Only participants with data available for specific study drug/metabolite were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 9
mcg | NA (NA) — Ae0-48 and fe0-48 of aleglitazar was not calculable (NC) since amount excreted in urine was below limit of quantification. | NA (NA) — Ae0-48 and fe0-48 of aleglitazar was not calculable (NC) since amount excreted in urine was below limit of quantification. | NA (NA) — Ae0-48 and fe0-48 of aleglitazar was not calculable (NC) since amount excreted in urine was below limit of quantification.

16. Secondary Outcome: Mean of Fraction of Unbound Aleglitazar (fu)
Description: fu was calculated using the mean of the 2-hour (reflecting Cmax) and 24-hour (reflecting Ctrough) values for each participant or, if the result of only one time-point was available, fu was the result of the available time-point. Ctrough) is a measured concentration at the end of a dosing interval at steady state.
Time Frame: 2 and 24 hours post-dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 6 | 7
Percentage | 0.101 (10.2) | 0.111 (7.4) | 0.114 (15.3)

17. Secondary Outcome: Area Under the Unbound Plasma Concentration-time Curve of Aleglitazar From Time 0 to Infinity (AUCu,Inf)
Description: AUCinf represents the area under the concentration-time curve of the analyte in plasma over the time interval from zero extrapolated to infinity. It was calculated by non-compartmental analysis using the linear trapezoidal rule, using relative actual time values. It was assessed using an analysis of variance model on the log-transformed values of AUCinf of aleglitazar with hepatic impairment group as factor.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 6 | 7
h*ng/mL | 0.0992 (27.0) | 0.122 (44.5) | 0.160 (30.0)
Statistical Analysis 1: Comparison: Normal Hepatic Function vs Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric Least-Squares Mean Ratio = 1.2323, 90% CI 2-sided [0.9618 to 1.5789]
Statistical Analysis 2: Comparison: Normal Hepatic Function vs Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Geometric Least-Squares Mean Ratio = 1.5587, 90% CI 2-sided [1.2165 to 1.9971]

18. Secondary Outcome: Maximum Unbound Plasma Concentration (Cmax,u) of Aleglitazar
Description: Cmax was obtained directly from the concentration-time data.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 6 | 7
ng/mL | 0.0213 (30.4) | 0.0214 (27.4) | 0.0257 (17.2)
Statistical Analysis 1: Comparison: Normal Hepatic Function vs Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric Least-Squares Mean Ratio = 1.0027, 90% CI 2-sided [0.8049 to 1.2492]
Statistical Analysis 2: Comparison: Normal Hepatic Function vs Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; GeometricLeast-Squares Mean Ratio = 1.2254, 90% CI 2-sided [0.9836 to 1.5266]

19. Secondary Outcome: Area Under the Unbound Plasma Concentration-time Curve of Aleglitazar From 0 to the Last Quantifiable Time-point Post-dose (AUCu,Last)
Description: Plasma samples were collected for this PK parameter. AUClast represents the area under the concentration-time curve of the analyte in plasma over the time interval from zero 0 to the last quantifiable time-point post-dose. It was calculated by non-compartmental analysis using the linear trapezoidal rule, using relative actual time values. AUClast was extrapolated to AUCinf by adding the ratio of Clast/kel to the AUClast, where Clast was the last observed concentration and kel was elimination rate constant.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 6 | 7
h*ng/mL | 0.0981 (27.3) | 0.121 (44.4) | 0.158 (29.6)

20. Secondary Outcome: Area Under the Unbound Plasma Concentration-time Curve of Aleglitazar From Time 0 to 48 Hours Post-dose (AUCu,0-48)
Description: AUClast represents the area under the concentration-time curve of the analyte in plasma over the time interval from zero to the 48 hours post-dose. It was calculated by non-compartmental analysis using the linear trapezoidal rule, using relative actual time values.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 15, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 6 | 7
h*ng/mL | 0.0980 (26.7) | 0.120 (40.9) | 0.158 (29.2)

21. Secondary Outcome: Apparent Unbound Volume of Distribution (Vz/Fu) of Aleglitazar
Description: VzF/u is an apparent volume of Unbound distribution during terminal phase after non-intravenous administration. It was calculated as CL/F/kel, where CL/F was calculated as dose/AUCinf, where AUCinf represents the area under the concentration-time curve of the analyte in plasma over the time interval from zero extrapolated to infinity and kel as constant elimination rate of aleglitazar.
Time Frame: as for outcome 9
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 6 | 7
L | 16600 (29.3) | 14500 (19.6) | 10600 (23.2)

22. Secondary Outcome: Apparent Unbound Total Body Clearance (CL/Fu) of Aleglitazar
Description: CL/F is an apparent total clearance of the drug from plasma after oral administration. It was calculated as dose/AUCinf. AUCinf represents the area under the concentration-time curve of the analyte in plasma over the time interval from zero extrapolated to infinity.
Time Frame: as for outcome 9
Population: The PK analysis population consisted of all participants who received the study drug and adhered to the protocol. Only participants with data available for specific study drug/metabolite were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 6 | 7
L/h | 1510 (27.0) | 1230 (44.5) | 939 (30.0)

23. Secondary Outcome: Number of Participants With Any Adverse Events (AEs), Serious Adverse Events (SAEs), Death, and Study Discontinuation
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect.
Time Frame: Up to 6 weeks
Population: The safety analysis consisted of all participants who had received the single dose of the study drug (aleglitazar), whether prematurely withdrawn from the study or not.
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
participants
  Any AEs | 3 | 0 | 2
  Any SAEs | 0 | 0 | 1
  Death | 0 | 0 | 0
  Study discontinuation | 0 | 0 | 1

24. Secondary Outcome: Number of Participants With Low and High Electrocardiograms (ECGs) Parameter Values
Description: The ECG evaluations were performed after participants were at rest and in supine position for at least 5 minutes before recording and remain resting and supine during the recordings. ECGs parameters included heart rate (HR), RR interval, PR interval, QRS duration, QT interval, QTcB, and QTcF intervals. The normal ranges of ECG parameter values were: HR as 40-100 beats per minute, RR as 600-1500 milliseconds (msec), PR as 120-200 msec, QRS as 80-120 msec, QT as 200-500 msec, QTcB as 350-450 msec, and QTcF as 350-450 msec. Data was reported as the number of participants who had low level values (values less than the normal range) and high level values (values more than the normal range).
Time Frame: Screening (Days -28 to -2), baseline (Day -1), Days 1 to 5, and follow-up visit (Day 10)
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
participants
  HR - high | 1 | 0 | 0
  HR - low | 0 | 0 | 0
  RR - high | 0 | 0 | 0
  RR - low | 1 | 0 | 0
  PR - high | 1 | 1 | 0
  PR - low | 2 | 0 | 3
  QRS - high | 0 | 0 | 0
  QRS - low | 6 | 1 | 6
  QT - high | 1 | 1 | 1
  QT - low | 0 | 0 | 0
  QTcB - high | 2 | 3 | 4
  QTcB - low | 0 | 0 | 0
  QTcF - high | 2 | 2 | 3
  QTcF - low | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Low and High Vital Signs Values
Description: Vital signs were assessed after participants had rested in a supine position for no less than 5 minutes. Vital signs included systolic blood pressure, diastolic blood pressure, pulse rate, and oral body temperature. The normal ranges of vital signs were: systolic blood pressure as 90-140 millimeter of Hg (mm Hg), diastolic blood pressure as 50-90 mm Hg, pulse rate as 45-100 beats per minute, and oral body temperature as 36.3-37.5 degree Celsius. Data was reported as the number of participants who had low level values (values less than the normal range) and high level values (values more than the normal range).
Time Frame: Days -28 to -2, Day -1, Days 1 to 5, and Day 10 for blood pressure and pulse rate; and Days -28 to -2, Day -1, and Day 10 for oral body temperature
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
participants
  Systolic blood pressure - high | 4 | 4 | 3
  Systolic blood pressure - low | 2 | 0 | 2
  Diastolic blood pressure - high | 2 | 3 | 1
  Diastolic blood pressure - low | 1 | 0 | 2
  Pulse rate - high | 1 | 0 | 0
  Pulse rate - low | 1 | 2 | 1
  Oral body temperature - high | 0 | 0 | 0
  Oral body temperature - low | 11 | 4 | 7

26. Secondary Outcome: Number of Participants With Marked Abnormalities in Clinical Laboratory Parameters
Description: Laboratory parameters included hematology, coagulation, biochemistry, and urinalysis. A marked abnormality was defined as a test result which was outside of the marked abnormality range. Data was reported as the number of participants who had low level values (values less than the normal range) and high level values (values more than the normal range).
Time Frame: Up to 6 weeks
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 18 | 10 | 10
participants
  Lymphocytes - low | 0 | 0 | 1
  Bicarbonate - high | 0 | 1 | 2
  Phosphate - high | 0 | 0 | 1
  Blood - high | 2 | 0 | 3
  Glucose - high | 0 | 0 | 3
  Protein - high | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Description: SAEs and other AEs were collected in the safety population, which was defined as all enrolled participants who received the single dose of the study drug, whether prematurely withdrawn from the study or not.
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 3/18 | 0/10 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Hepatic Function (N=18) | Mild Hepatic Impairment (N=10) | Moderate Hepatic Impairment (N=10)
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Hepatic Function (N=18) | Mild Hepatic Impairment (N=10) | Moderate Hepatic Impairment (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Nasal decongestion therapy (Surgical and medical procedures) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.